CLINICAL TRIAL: NCT06888713
Title: Telemonitoring of Activities of Daily Living in Home Care Services of Older Adults with Cognitive Deficits: a Large-scale Action Design Research Study
Brief Title: Telemonitoring of Activities of Daily Living in Home Care Services of Older Adults with Cognitive Deficits
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Principal Investigator, Nathalie Bier, Full professor, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PJT-195697
Record Dates: First submitted 2025-02-28; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Dementia
Keywords: Telemonitoring of ADL; Homecare services; IA
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemonitoring of ADL group (Experimental): Will receive the technology in their home to document if it influenced the homecare services plan.
  Interventions: Other: Telemonitoring of ADL
- No telemonitoring of ADL (No Intervention): Another group will be followed in therms of homecare services received, but without the technology. The control group will be gathered based on archives data only.

INTERVENTIONS:
Other: Telemonitoring of ADL — Telemonitoring of ADL is based on smart environments sensors (non wearables) and gathers information about activity of daily living routines for a better understanding of homecare services needed.
  Arms: Telemonitoring of ADL group

SUMMARY:
In Canada, it is estimated that two million people are users of publicly funded home care services, with more than half of them being 65 years and older. Although home care services are considered a priority by Canadian provinces, in Québec alone, more than 46 000 people were waiting for those services in 2022. The provision of home care services is hampered by limited funding and growing demand from among an aging population, among other factors. These challenges have led to urgent calls to better support home care in Canada to ensure optimal use of scarce human and financial resources. One of the key strategies to achieve optimal use of resources may be remote monitoring of activities of daily living (ADLs), a type of telehealth. ADL telemonitoring can remotely recognize ADLs such as preparing meals and moving around the home. Past studies have shown that ADL telemonitoring can help in better understanding older adults' home care needs, thereby allowing for more personalized ADL interventions. Previous projects have also allowed for the developement of NEARS-SAPA, a telemonitoring system for ADLs. In these past projects, it was identified how NEARS-SAPA was used by home care services and its ease of use was tested in real environments. In the present project, the benefits of ADL telemonitoring will be tested and its technological capabilities expanded, hence preparing the system for the next big step, i.e. large-scale adoption by home care services. Ultimately, ADL telemonitoring may help the healthcare system determine which service is more appropriate for which person and at what time, thereby optimizing interventions and resource management.

ELIGIBILITY:
Inclusion Criteria:

1) be an older adult (> 65 years old), 2) have cognitive deficits as reported in the medical record, 3) live alone, at home, 4) be a care recipient of home care services, 5) speak French or English

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of homecare services received to support activities of daily living (ADL) | From enrollment until around 12 months of following.
  Number of homecares ADL services received as identified in clinical databases.
Nature of homecare services received to support activities of daily living (ADL). | From enrollement until around 12 months of following.
  The category of services received related to ADL as indicated in clinical databases.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Bier, Ph.D., Principal Investigator — CRIUGM, Université de Montréal; Charles Gouin-Vallerand, Ph.D., Principal Investigator — Université de Sherbrooke; Kevin Bouchard, Ph.D., Principal Investigator — Université du Québec à Chicoutimi

IPD SHARING:
Plan to Share IPD: Undecided